CLINICAL TRIAL: NCT00197652
Title: Botswana Diarrheal Diseases Study
Status: Completed | Type: Observational
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Botswana Ministry of Health (Other Government)
Responsible Party: Principal Investigator, Roger Shapiro, Principal Investigator, Harvard School of Public Health (HSPH)
Other Study IDs: K23HD001330-05 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2011-10-07 (Estimated); Status verified 2011-10

CONDITIONS: HIV Infections
Keywords: Prevention of Mother-Infant HIV Transmission
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Diarrheal specimens from infants born to HIV infected mothers: 400 diarrheal specimens will suffice to determine the prevalence of specific pathogens in the region. Of these, 300 specimens will be collected from infants born to HIV infected mothers, and 100 specimens will be collected from infants born to HIV uninfected mothers.
- Breast milk from HIV infected and HIV uninfected women: Breast milk from HIV infected and HIV uninfected women who are breastfeeding is collected at 2 days, 2 weeks, 2 months, and 5 months post-partum. This breast milk will be compared for in vitro functional quality of immunoglobulins to selected diarrheal and respiratory pathogens.

SUMMARY:
The goals of this study are to:

1. determine the diarrheal rates, morbidity, mortality, and pathogens present among breast-fed infants born to HIV-infected mothers.

   * analysis by HIV status of infants, method of feeding, HIV viral loads / CD4 counts of infected mothers.
   * comparison to rates among infants born to HIV uninfected mothers.
2. link analysis of the functional quality of immunoglobulins in the breast milk of HIV-infected and uninfected mothers.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to provide independent informed consent.
* Subject is able to complete a questionnaire as part of her enrollment visit and agrees to complete follow-up questionnaires monthly.
* Subject presents symptoms of acute diarrhea: at least 3 loose stools during 24 hours as reported by mother; persistent diarrhea: an episode of diarrhea lasting 14 days; recurrent diarrhea: a new episode of diarrhea after an interval of at least two diarrhea-free days.

For HIV-infected subjects:

* Mother: HIV antibody is detected by dual HIV-1 ELISA and confirmed by western blot. Infant: HIV antigen is detected by PCR on 2 samples during the follow-up period, or on 1 sample followed by the death of the infant.

Exclusion Criteria:

* Subject cannot provide legal independent informed consent.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 1350 (Actual)
Dates: Start 2001-03; Primary Completion 2003-10 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
OCCURRENCE OF SUSPECTED PNEUMONIA OR BLOODSTREAM INFECTION OVER FIRST TWO YEARS OF LIFE | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Roger Shapiro, MD, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- Princess Marina Hospital, Gaborone, Botswana

REFERENCES:
- [Derived] Shapiro RL, Smeaton L, Lockman S, Thior I, Rossenkhan R, Wester C, Stevens L, Moffat C, Arimi P, Ndase P, Asmelash A, Leidner J, Novitsky V, Makhema J, Essex M. Risk factors for early and late transmission of HIV via breast-feeding among infants born to HIV-infected women in a randomized clinical trial in Botswana. J Infect Dis. 2009 Feb 1;199(3):414-8. doi: 10.1086/596034. PMID 19090775
- [Derived] Shapiro RL, Lockman S, Kim S, Smeaton L, Rahkola JT, Thior I, Wester C, Moffat C, Arimi P, Ndase P, Asmelash A, Stevens L, Montano M, Makhema J, Essex M, Janoff EN. Infant morbidity, mortality, and breast milk immunologic profiles among breast-feeding HIV-infected and HIV-uninfected women in Botswana. J Infect Dis. 2007 Aug 15;196(4):562-9. doi: 10.1086/519847. Epub 2007 Jul 9. PMID 17624842